CLINICAL TRIAL: NCT00164320
Title: Project TEAM: Teaching HIV Prevention in the HIV Clinic
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: CDC-NCHSTP-3699; R18/CCR420971-01
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2005-09-14 (Estimated); Status verified 2005-09

CONDITIONS: HIV

INTERVENTIONS:
Behavioral: TEAM

SUMMARY:
The purpose of this study is to determine if the TEAM prevention intervention delivered by a physician and an HIV-positive counselor is effective. It is hypothesized that those who receive the intervention will report a higher reduction in risky sex than those who were in the standard-care condition.

ELIGIBILITY:
Inclusion Criteria:

* 1) 18 years or older, 2) HIV-infected, 3) Sexually active, 3)Receiving HIV primary care at participating clinic, 4) Can communicate in English or Spanish, 5) No previous enrollment in the TEAM study or intervention.

Exclusion Criteria:

* 1) Participation in a similar study run by the TEAM PI.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 600
Dates: Start 2004-05; Study Completion 2006-05

PRIMARY OUTCOMES:
Self-reported unprotected (without condoms)anal or vaginal sex with HIV-negative or unknown-status persons.

CONTACTS AND LOCATIONS:
Overall Officials: Dogan Eroglu, PhD., Study Director — Centers for Disease Control and Prevention; Lisa Metsch, PhD., Principal Investigator — University of Miami
Locations (1):
- University of Miami School of Medicine, Miami, Florida, United States